CLINICAL TRIAL: NCT04280952
Title: Confocal Laser Endomicroscopy for Brain Tumors
Acronym: CONVIVO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CONVIVO
Record Dates: First submitted 2020-02-20; First posted 2020-02-21 (Actual); Last update posted 2023-07-05 (Actual); Status verified 2023-07

CONDITIONS: Brain Tumor; Surgery; Convivo System; Laser Endomicroscopy
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Intervention Model Description: Tumor tissue identification with CONVIVO system
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CONVIVO (Experimental): tumor tissue identification with the CONVIVO system
  Interventions: Device: CONVIVO

INTERVENTIONS:
Device: CONVIVO — tumor tissue with the CONVIVO system

SUMMARY:
The prognosis of glioblastoma patients highly depends on resection extent. Various strategies have been introduced to overcome the dilemma of intraoperative tumor identification.

In gastroenterology, confocal laser endomicroscopy (CLE) allows precise differentiation of tumor tissue from surrounding mucosa in various diseases. Combining high-definition white light endoscopy with CLE significantly increases sensitivity and specificity compared with the sole application of high-definition white light endoscopy.

CLE was recently introduced to neurosurgical applications. Although still in an early stage of clinical application, this technique has proven to be capable of differentiating various tumor entities in animal models as well as human tissue samples. CLE allows visualization of the underlying tissue on a microscopic scale, receiving information on the microstructure as well as cellular components. However, the clinical importance of this technique for its application in neurosurgery will be demonstrated in this clinical trial.

DETAILED DESCRIPTION:
Background:

The prognosis of glioblastoma patients highly depends on resection extent. Various strategies have been introduced to overcome the dilemma of intraoperative tumor identification.

In gastroenterology, confocal laser endomicroscopy (CLE) allows precise differentiation of tumor tissue from surrounding mucosa in various diseases. Combining high-definition white light endoscopy with CLE significantly increases sensitivity and specificity compared with the sole application of high-definition white light endoscopy.

CLE was recently introduced to neurosurgical applications. Although still in an early stage of clinical application, this technique has proven to be capable of differentiating various tumor entities in animal models as well as human tissue samples. CLE allows visualization of the underlying tissue on a microscopic scale, receiving information on the microstructure as well as cellular components. However, the clinical importance of this technique for its application in neurosurgery still needs to be demonstrated

Methods:

Intravenous injection dose of fluorescein sodium. For every operation the investigators plan to take pictures with the CONVIVO system before taking the material for standard frozen section and definitive histopathology. These pictures will be evaluated by a pathologist afterwards.

Objectives:

The primary objective of this trial is to demonstrate, that the CONVIVO system allows identification of tumor tissue. The secondary objectives are procedural aspects and handling issues covering the usability.

ELIGIBILITY:
Inclusion Criteria:

* The patient is undergoing neurosurgery for a suspected brain tumor and amenable to surgical resection by fluorescent guided technique
* The patient has an indication for tumor resection
* Macroscopic tumor visualization using sodium fluorescein is planned, concentration 5-10mg/kg
* The patient is older than 18 years
* Written consent

Exclusion Criteria:

* Stereotactic biopsy procedure
* Patients with any kind of contraindication to the use of fluorescein sodium
* Vulnerable persons (pregnant women, patients with Glasgow Coma Scale below 14)
* Participation in other ongoing clinical trials with one exception: double inclusions are allowed provided that no interaction with NaF is to be expected
* People who do not want to participate in the study
* Tumors that do not exactly match the inclusion criteria
* Emergency procedures in which no consent was obtained before the operation.
* Multiple surgeries on the same patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2020-06-05 (Actual); Primary Completion 2023-06-13 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Identification of tumor tissue | End of surgery
  Identification of tumor tissue versus non-affected tissue by the CONVIVO system in comparison to the histopathology of frozen section

SECONDARY OUTCOMES:
Accuracy of CONVIVO results | 14 days after surgery
  Accuracy of CONVIVO results compared with results of final tumor histopathology
Time for tissue visualization with the CONVIVO system | End of surgery
  Intraoperative time for the tissue visualization with the CONVIVO system
Rate of unclear visualizations | 14 days after surgery
  Rate of unclear visualizations in %

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Seidel, MD, Principal Investigator — Principal Investigator
Locations (1):
- Dep. of Neurosurgery, Bern University Hospital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No